CLINICAL TRIAL: NCT01945879
Title: Pilot Study of Intensified Chemotherapy and Simultaneous Treatment With Heparin in Out-patients With Pancreatic Cancer.
Brief Title: Pilot Safety Trial of Chemotherapy and Use of Heparin in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CONKO-Studiengruppe (Other)
Responsible Party: Principal Investigator, Uwe Pelzer MD, MD, CONKO-Studiengruppe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONKO-004/1
Record Dates: First submitted 2013-09-05; First posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; heparin; thromboembolic events; bleedings
MeSH Terms: conditions — Pancreatic Neoplasms; Thromboembolism | interventions — Enoxaparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GFFC + LMWH (Experimental): gemcitabine/ 5-flourouracil/folinic acid/ cisplatin as chemotherapeutic treatment plus enoxaparine as experimental addition
  Interventions: Drug: Enoxaparine

INTERVENTIONS:
Drug: Enoxaparine — al patients received additional low molecular heparin, if the safety cohort of three patients received at least 4 weeks of combined treatment without severe side effects, recruitment were continued until a minimum of 15 patients completed at least 3 months of treatment.
  Other Names: low molecular weight heparin; clexane

SUMMARY:
Venous thromboembolic events are considered to be a prognostic negative factor and small studies showed astonishing survival advantages using heparin as prophylactic treatment to prevent venous thromboembolic events. Based on these assumptions our Charité - Onkologie (CONKO) study group planned to conduct a randomized trial to investigate the impact of low molecular weight heparin (LMWH) in a prospective setting in patients with advanced pancreatic cancer undergoing first line therapy, the CONKO-004 trial. During the preliminary stages we had to undertake a pilot trial to get information on safety and feasibility of combined chemotherapy with simultaneous treatment of the LMWH Enoxaparin in patients with advanced pancreatic cancer who are at high risk of gastrointestinal bleeding due to local cancer spread.

DETAILED DESCRIPTION:
The trial was a prospective, open-label, single center investigation in patients with inoperable pancreatic cancer who were treated with first-line chemotherapy in an outpatient setting. The intensified treatment consisted of gemcitabine 1g/m² (30 min), 5-flourouracil 750 mg/m² (24 h), folinic acid 200 mg/m² (30 min), and Cisplatin 30 mg/m² (90 min) on day 1 and 8; q3w). Beyond initial 3 months of intensified chemotherapy all patients without cancer progression received further treatment with gemcitabine alone to prevent patients from cumulative toxicities. The concomitant use of Enoxaparin started on day 1 of chemotherapy with a fixed dose of 40 mg daily until cancer progression. Dose adjustment for enoxaparin was recommended in patients with impaired kidney function or thrombocytopenia within the study according to National Cancer Institute Common Toxicity Criteria guidelines to minimize bleeding risk. Prophylactic antiemetic therapy and supportive care were provided according to individual symptoms and demand.

The study used a sequential design to be able to stop the feasibility investigation in case of severe side effects. After inclusion of three consecutive patients a hold of recruitment was arranged until all three patients received at least 4 weeks of concomitant enoxaparin treatment. In absence of serious events the recruitment should be continued until a minimum of 15 patients received at least 12 weeks concomitant enoxaparin treatment.

The trial was approved by the Scientific and Research Ethics Committee of our institution. The investigation was conducted in accordance with the Declaration of Helsinki and Good Clinical Practice Guidelines. Furthermore, the national principles for the proper execution of the clinical examination of drugs ("Bundesanzeiger" No. 243 of 30.12.1987), the national regulations of the German drug law, and the German drug test guidelines were adhered.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory patients with histologically confirmed advanced adenocarcinoma of the pancreas
* no previous radio- or chemotherapy
* Karnofsky Performance Status (KPS) ≥ 60%
* measurable tumour lesion confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) within the last 14 days
* no VTE within the last 2 years
* adequate compliance and home residence within geographical proximity to the particular department (allowing an adequate follow-up)
* sufficient bone marrow function (leukocytes 3.5 × 109/l, thrombocytes 100 × 109/l)
* age ≥ 18 years.

Exclusion Criteria:

* pre-existing indication for anticoagulation
* major bleeding events within the last 2 weeks
* severe impairment of coagulation
* active gastrointestinal ulcers or major surgery within the last 2 weeks
* body weight < 45kg or > 100kg
* pregnancy/lactation or insufficient contraception during study
* severely impaired renal function (creatinine clearance < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-01; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Incidence of NCI CTC Toxicity III°/IV° and severe bleedings | minimum of 3 months
  Incidence of NCI CTC Toxicity III°/IV° as well as severe bleedings for a minimum of 15 patients and an observation time of at least 3 months

SECONDARY OUTCOMES:
overall survival | at least 12 months of follow up
  Secondary aims were overall survival (OS), the impact of patients characteristics on survival and the rate of symptomatic venous thromboembolic events and major bleedings

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Pelzer, MD, Principal Investigator — Charité - Universitaetsmedizin Berlin
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Pelzer U, Hilbig A, Stieler JM, Bahra M, Sinn M, Gebauer B, Dorken B, Riess H. Intensified chemotherapy and simultaneous treatment with heparin in outpatients with pancreatic cancer - the CONKO 004 pilot trial. BMC Cancer. 2014 Mar 19;14:204. doi: 10.1186/1471-2407-14-204. PMID 24641937